CLINICAL TRIAL: NCT05435768
Title: PhaseⅠ-Ⅱ Clinical Study of Hypofractionated Radiotherapy Combined With PD-1 Inhibitor Sequential GM-CSF(PraG) With RANKL Inhibitor for the Treatment of Advanced Multiple Metastatic Solid Tumors
Brief Title: PraG With RANKL Inhibitor for the Treatment of Advanced Multiple Metastatic Solid Tumors
Acronym: PRaG 2X
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-LK-2022-035-01
Record Dates: First submitted 2022-06-12; First posted 2022-06-28 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A :RANKL inhibitor subsequently HFRT+GM-CSF+PD-1 inhibitor: Group A(6 patients):patients were subcutaneously injected with 120mg desomumab, and on the second day after injection, the metastatic lesions were treated with hypofractioniated radiotherapy (8Gy×3F or 5Gy×3F), and subcutaneously injected with GM-CSF(200 μg/d) for 7 days, followed by IL-2 (2 million IU/d) for 7 days,and a 200mg PD-1 inhibitor administered within one week after completion of radiotherapy. The course was repeated every 28 days for 2-4 cycles.After combination therapy, maintenance therapy with PD-1inhibitor and desomumab was administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Denosumab
- Group B:HFRT+GM-CSF+PD-1 inhibitor subsequently RANKL inhibitor: Group B(6 patients):patients were treated with hypofractioniated radiotherapy (8Gy×3F or 5Gy×3F), and subcutaneously injected with GM-CSF(200 μg/d) for 7 days, followed by IL-2 (2 million IU/d) for 7 days.On the second day after radiotherapy, 200mg pd-1 inhibitor was administered. After treatment, 120mg desomumab was subcutaneously injected. The course was repeated every 28 days for 2-4 cycles.After combination therapy, maintenance therapy with PD-1inhibitor and desomumab was administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab 120mg was subcutaneously administered one day before the commencement of radiotherapy or after the PraG treatment every 28 days

SUMMARY:
The PraG treatment model has synergistic effects with RANKL inhibitor therapy, and the combination of the two treatments provides a survival benefit for patients with multiple bone metastatic solid tumors who have failed first-line systemic therapy. Phase I clinical trial is planned to determine the safety of PraG treatment mode combined with RANKL inhibitor desomumab and the optimal treatment sequence and mode. Further phase II clinical trial was conducted to confirm the efficacy of PraG treatment combined with desomumab. The mechanism of combination therapy was analyzed and biomolecular markers for potential efficacy prediction were screened by detection of lymphocyte subsets, cytokines and metabolomics in peripheral blood.

DETAILED DESCRIPTION:
Group A(6 patients):patients were subcutaneously injected with 120mg desomumab, and on the second day after injection, the metastatic lesions were treated with hypofractioniated radiotherapy (8Gy×3F or 5Gy×3F), and subcutaneously injected with GM-CSF(200 μg/d) for 7 days, followed by IL-2 (2 million IU/d) for 7 days,and a 200mg PD-1 inhibitor administered within one week after completion of radiotherapy. The course was repeated every 28 days for 2-4 cycles.After combination therapy, maintenance therapy with PD-1inhibitor and desomumab was administered until disease progression or unacceptable toxicity.

Group B(6 patients):patients were treated with hypofractioniated radiotherapy (8Gy×3F or 5Gy×3F), and subcutaneously injected with GM-CSF(200 μg/d) for 7 days, followed by IL-2 (2 million IU/d) for 7 days.On the second day after radiotherapy, 200mg pd-1 inhibitor was administered. After treatment, 120mg desomumab was subcutaneously injected. The course was repeated every 28 days for 2-4 cycles.After combination therapy, maintenance therapy with PD-1inhibitor and desomumab was administered until disease progression or unacceptable toxicity.

The phase II study followed the treatment modality of the cohort with higher safety and efficacy assessments in the Phase I study and additional 39 patients were added.The primary endpoint is disease control rate. Secondary endpoints were objective response rate (ORR), median progression-free survival (PFS), overall survival (OS), and incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years
2. The patients must conform to the advanced solid cancer with multiple metastases(may be accompanied by metastasis of other organs),progression after first-line systemic therapy and have clear pathological diagnosis report
3. The hematopoietic function and general condition of the patients were acceptable(white blood cells >2.5×10^9/L,lymphocyte>0.5 times of normal lower limit，Platelets>50×10^9/L）
4. There was no history of serious hematopoietic function, abnormal heart, lung, liver, kidney function and immune deficiency
5. One week before enrollment,absolute value of T lymphocytes≥0.5 times of normal lower limit，neutrophil ≥ 1.0×109/L，AST and ALT ≤3.0 times normal upper limit(Liver cancer/liver metastasis patients ≤5.0 times normal upper limit);creatinine ≤ 3.0 times normal upper limit;serum calcium≥2.0mmol/L
6. Patients's activity status was assessed by Eastern Cooperative Oncology Group(ECOG) score of 0-3,and life expectancy of more than 3 months
7. Abide by the plan during the study period
8. Sign written consent

Exclusion Criteria:

1. Pregnant or lactating women
2. Patinets diagnosed with other malignant disease in the past five years,except for cured skin cancer and cervical carcinoma in situ
3. The clinical severity of uncontrolled epilepsy,central nervous system disease or mental disorder may hinder the signing of informed consent or affect the patient's compliance with medication
4. Sever(i.e. active)heart disease,such an symptomatic coronary heart disease,New York Heart Association(NYHA) class Ⅱ or more severe congestive heart failure or severe arrhythmia requiring drug intervention,or a history of myocardial infraction in the last 12 months；
5. Organ transplantation require immunosuppressive therapy
6. Major active infections are known,or other serious uncontrolled concomitant diseases;endocrine or metabolic disorders,or other serious uncontrolled concomitant diseases;
7. The baseline blood routine did not meet the following criteria:hemoglobin≥90g/L;absolute neutrophil count(ANC)≥1.5×109/L;platelet≥50×109/L;ALT,AST≤2.5 times normal upper limit value;ALP≤2.5 times normal upper limit value; serum total bilirubin<1.5 times normal upper limit value;Serum creatinine <3 times normal upper limit value;serum albumin≥30g/L;
8. Anaphylaxis to any research drug ingredients
9. Patients with a history of immunodeficiency,including HIV postive or with other acquired or congenital immunodeficiency disorders,or with a history of organ transplantation,or with other immune-related diseases requiring long-term oral hormone therapy
10. In the period of acute and chronic tuberculosis infection (T-spot test positive,chest X-ray suspicious tuberculosis focus patients)
11. Researchers considered that it was not suitable for other situations in the group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced solid tumors with multiple bone metastases
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2022-08-16 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Does limiting toxicity（CTC 5.0） | phase 1 (1 year)
DCR | phase 2 (18 months)
  CR+PR+SD(RECIST 1.1)

SECONDARY OUTCOMES:
objective response rate | after 12-weeks treatment
progression-free survival | after 12-weeks treatment
overall survival | after 12-weeks treatment
incidence of skeletal related events | phase 1/2 (30 months)
toxic response | phase 2 (18 months)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Result] Kong Y, Ma Y, Zhao X, Pan J, Xu Z, Zhang L. Optimizing the Treatment Schedule of Radiotherapy Combined With Anti-PD-1/PD-L1 Immunotherapy in Metastatic Cancers. Front Oncol. 2021 Mar 30;11:638873. doi: 10.3389/fonc.2021.638873. eCollection 2021. PMID 33859942
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33859942/